CLINICAL TRIAL: NCT03743324
Title: A Multi-center Prospective Observational Trial Investigating the Effect of Radiation and Its Timing on Breast Reconstruction in Chinese Patients
Brief Title: Effect of Radiation and Its Timing on Breast Reconstruction in Chinese Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E2018210
Record Dates: First submitted 2018-11-07; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: breast reconstruction; Chinese; radiation; timing
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BR group: Breast reconstruction without radiation therapy
  Interventions: Procedure: Immediate Breast reconstruction; Procedure: Delayed Breast Reconstruction
- Immediate BR +post-op radiation: Immediate breast reconstruction followed by surgical site radiation therapy
  Interventions: Procedure: Immediate Breast reconstruction; Radiation: Radiation
- Radiation +delayed BR: previous post-mastectomy radiation followed by delayed breast reconstruction
  Interventions: Procedure: Delayed Breast Reconstruction; Radiation: Radiation

INTERVENTIONS:
Procedure: Immediate Breast reconstruction — Immediate Autologous/prosthetic-based breast reconstruction is performed after mastectomy on the breast that is diagnosed with breast cancer
  Groups: BR group; Immediate BR +post-op radiation
Procedure: Delayed Breast Reconstruction — Delayed Autologous/prosthetic-based breast reconstruction is performed after mastectomy on the breast that is diagnosed with breast cancer
  Groups: BR group; Radiation +delayed BR
Radiation: Radiation — Radiation is performed to the surgical site and complies with the ASCO guidelines on post-mastectomy radiotherapy
  Groups: Immediate BR +post-op radiation; Radiation +delayed BR

SUMMARY:
The purpose of the study is to investigate the impacts of radiation and the timing of radiation on autologous and prosthetic-based breast reconstruction in Chinese post-mastectomy breast cancer patients. The study aims to optimize the timing for autologous/prosthetic breast reconstruction which delivers the best aesthetic results while maintains low complication rate and best integrates into the comprehensive breast cancer treatment. The study is open to all female breast cancer patients undergoing breast reconstruction in the department of breast reconstruction in Tianjin medical university cancer institute and hospital.

DETAILED DESCRIPTION:
In breast cancer patients, post-operative radiation therapy is an important component in breast cancer management. However, in the context of breast reconstruction, radiation can have adverse effect as it increases the rate of fat necrosis and leads to fibrosis/ capsular contracture in the reconstructed breast mounds. It is therefore necessary to investigate the best timing for breast reconstruction, especially in those patients which post-operative radiation is required, which does not interfere with overall breast cancer treatment while produces the best surgical, aesthetic and psychological outcome. Most studies in this field are retrospective, and studies on Chinese cohort are also rare. This multi-center prospectively designed clinical trial will include several medical centers across China. The investigators will allocate the patients into three arms based on the status and sequence of radiation and breast reconstruction, and will further stratify the groups based on the different approaches of reconstruction (autologous/ prosthetic based). Both objective and subjective (patient oriented) methods will be employed to make evaluations involving surgical, aesthetic, and psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer
* Karnofsky Performance Status (KPS) larger than 70
* Underwent autologous or prosthetic based breast reconstruction
* No severe deficiency in hematological, cardiovascular system, no immune-deficiency, no severe abnormal liver or kidney function.

Exclusion Criteria:

* Metastatic breast cancer
* Local recurrence after mastectomy
* Prior radiation history to chest wall due to other tumors
* Radiation performed more than 6 months after mastectomy
* Interruption of radiation more than 2 weeks
* Gravida or during lactation
* Concurrently undergoing psychotic disorders

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female breast patients who have natural breasts
Study Population: Study population include female Chinese breast cancer patients who wish to undergo autologous or prosthetic-based breast reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 1344 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
occurrence of short term complications | the short term complications will be inspected up to 3 months post-op;
  impaired arterial or venous flap perfusion by increased (>3 seconds) or reduced (<2 seconds) capillary refill time; infection of the reconstructed breast with evidences from microbiological cultures; partial or entire flap necrosis with evident demarcation by clinical observation
occurrence and change of long term complications | the long term complications will be assessed at 6 months post-op; repeated assessments will be made at 12 and 24 months to record changes
  fat necrosis proven by breast ultrasound/ breast MRI/ pathology; flap contracture that causes change in shape and/or volume in the reconstructed breast mound observed by naked-eye inspection or breast imaging; capsular contracture that causes hardness/pains or changes of the reconstructed breast mound observed by surgeon's inspection or breast imaging.
occurrence of secondary surgery | up to 24 months post-op
  unplanned surgery due to short-term and/or long-term complications post-op, the types of secondary surgery include but not limited to exploratory surgery, flap salvages, removal or fat necrosis, debridement, prosthetic explantation.

SECONDARY OUTCOMES:
occurrence of revision surgery | 6 to 24 months post-op
  any surgery performed to the reconstructed or contralateral breast to optimize symmetry
baseline and change of subjective evaluation | the baseline evaluation will be made at 6 months post-op; repeated evaluations will be made at 12 and 24 months to record changes
  patient oriented aesthetic, psychological and overall outcome evaluations are made with BREAST-Q (short for breast-questionnaire) post reconstruction module, the the selected questionnaire includes a set of questions regarding : category 1-patients' satisfaction with breasts; category 2-patients' satisfaction with outcome and category 3-patients' psychological well-being. In each category, the total score is generated by Q-score (short for questionnaire-score)software and the total score ranges from 0-100. The higher the score the better the satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yin, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Background] Schaverien MV, Macmillan RD, McCulley SJ. Is immediate autologous breast reconstruction with postoperative radiotherapy good practice?: a systematic review of the literature. J Plast Reconstr Aesthet Surg. 2013 Dec;66(12):1637-51. doi: 10.1016/j.bjps.2013.06.059. Epub 2013 Jul 22. PMID 23886555
- [Background] Berbers J, van Baardwijk A, Houben R, Heuts E, Smidt M, Keymeulen K, Bessems M, Tuinder S, Boersma LJ. 'Reconstruction: before or after postmastectomy radiotherapy?' A systematic review of the literature. Eur J Cancer. 2014 Nov;50(16):2752-62. doi: 10.1016/j.ejca.2014.07.023. Epub 2014 Aug 26. PMID 25168640
- [Background] Barry M, Kell MR. Radiotherapy and breast reconstruction: a meta-analysis. Breast Cancer Res Treat. 2011 May;127(1):15-22. doi: 10.1007/s10549-011-1401-x. Epub 2011 Feb 20. PMID 21336948
- [Background] Kelley BP, Ahmed R, Kidwell KM, Kozlow JH, Chung KC, Momoh AO. A systematic review of morbidity associated with autologous breast reconstruction before and after exposure to radiotherapy: are current practices ideal? Ann Surg Oncol. 2014 May;21(5):1732-8. doi: 10.1245/s10434-014-3494-z. Epub 2014 Jan 29. PMID 24473643
- [Background] Losken A, Nicholas CS, Pinell XA, Carlson GW. Outcomes evaluation following bilateral breast reconstruction using latissimus dorsi myocutaneous flaps. Ann Plast Surg. 2010 Jul;65(1):17-22. doi: 10.1097/SAP.0b013e3181bda349. PMID 20548235
- [Background] Selber JC, Kurichi JE, Vega SJ, Sonnad SS, Serletti JM. Risk factors and complications in free TRAM flap breast reconstruction. Ann Plast Surg. 2006 May;56(5):492-7. doi: 10.1097/01.sap.0000210180.72721.4a. PMID 16641623
- [Background] Chang EI, Liu TS, Festekjian JH, Da Lio AL, Crisera CA. Effects of radiation therapy for breast cancer based on type of free flap reconstruction. Plast Reconstr Surg. 2013 Jan;131(1):1e-8e. doi: 10.1097/PRS.0b013e3182729d33. PMID 23271550
- [Background] Kronowitz SJ. Current status of implant-based breast reconstruction in patients receiving postmastectomy radiation therapy. Plast Reconstr Surg. 2012 Oct;130(4):513e-523e. doi: 10.1097/PRS.0b013e318262f059. PMID 23018711
- [Background] Pestana IA, Campbell DC, Bharti G, Thompson JT. Factors affecting complications in radiated breast reconstruction. Ann Plast Surg. 2013 May;70(5):542-5. doi: 10.1097/SAP.0b013e31827eacff. PMID 23542851
- [Background] Chatterjee JS, Lee A, Anderson W, Baker L, Stevenson JH, Dewar JA, Thompson AM. Effect of postoperative radiotherapy on autologous deep inferior epigastric perforator flap volume after immediate breast reconstruction. Br J Surg. 2009 Oct;96(10):1135-40. doi: 10.1002/bjs.6693. PMID 19787763
- [Background] Rogers NE, Allen RJ. Radiation effects on breast reconstruction with the deep inferior epigastric perforator flap. Plast Reconstr Surg. 2002 May;109(6):1919-24; discussion 1925-6. doi: 10.1097/00006534-200205000-00022. PMID 11994594
- [Background] Yueh JH, Slavin SA, Adesiyun T, Nyame TT, Gautam S, Morris DJ, Tobias AM, Lee BT. Patient satisfaction in postmastectomy breast reconstruction: a comparative evaluation of DIEP, TRAM, latissimus flap, and implant techniques. Plast Reconstr Surg. 2010 Jun;125(6):1585-1595. doi: 10.1097/PRS.0b013e3181cb6351. PMID 20517080
- [Background] Lam TC, Hsieh F, Boyages J. The effects of postmastectomy adjuvant radiotherapy on immediate two-stage prosthetic breast reconstruction: a systematic review. Plast Reconstr Surg. 2013 Sep;132(3):511-518. doi: 10.1097/PRS.0b013e31829acc41. PMID 23676964
- [Background] He S, Yin J, Robb GL, Sun J, Zhang X, Li H, Liu J, Han C. Considering the Optimal Timing of Breast Reconstruction With Abdominal Flaps With Adjuvant Irradiation in 370 Consecutive Pedicled Transverse Rectus Abdominis Myocutaneous Flap and Free Deep Inferior Epigastric Perforator Flap Performed in a Chinese Oncology Center: Is There a Significant Difference Between Immediate and Delayed? Ann Plast Surg. 2017 Jun;78(6):633-640. doi: 10.1097/SAP.0000000000000927. PMID 27798424